CLINICAL TRIAL: NCT02306109
Title: Effects of Motor Rehabilitation Treatment on Disability and Quality of Life in Amyotrophic Lateral Sclerosis (ALS).
Brief Title: Effect of Motor Rehabilitation Treatment on Amyotrophic Lateral Sclerosis (ALS)
Acronym: ermoSla
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Unita' Sanitaria Locale Di Modena (Other)
Collaborators: University of Modena and Reggio Emilia (Other); Azienda USL Reggio Emilia - IRCCS (Other Government); S. Anna Hospital (Other); Azienda Unità Sanitaria Locale Ferrara (Unknown)
Responsible Party: Principal Investigator, Jessica Mandrioli, MD, Department of Neuroscience, St. Agostino-Estense Hospital, Modena (IT), Azienda Unita' Sanitaria Locale Di Modena
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AUSLMO_0001_SLA
Record Dates: First submitted 2014-11-21; First posted 2014-12-03 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Motor Rehabilitation Treatment; Intensive versus standard; Motor Disability
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard motor rehabilitation treatment (Active Comparator)
  Interventions: Procedure: Standard motor rehabilitation treatment
- Intensive motor rehabilitation treatment (Experimental)
  Interventions: Procedure: Intensive motor rehabilitation treatment

INTERVENTIONS:
Procedure: Standard motor rehabilitation treatment — Standard treatment: 2 sessions/week of motor rehabilitation treatment (45 minutes each one) for 10 weeks for a total of 20 sessions, including exercises for aerobic endurance, reinforcement at low load and stretching. At the end of the 20 sessions, patient and caregiver are going to continue motor activity with therapist supervision through regular follow up
  Arms: Standard motor rehabilitation treatment
Procedure: Intensive motor rehabilitation treatment — Intensive treatment is characterized by an increased exercises volume: 5 sessions/week)(45 minutes each one) for 10 weeks for a total of 50 sessions, including exercises for aerobic endurance, reinforcement at low load and stretching. At the end of the 50 sessions, patient and caregiver are going to continue motor activity with therapist supervision through regular follow up
  Arms: Intensive motor rehabilitation treatment

SUMMARY:
ErmoSLA is a multicentric, randomized, controlled trial to compare effects of an "intensive" or "standard" motor rehabilitation treatment on motor disability in people with ALS

DETAILED DESCRIPTION:
The study is a multicentric, randomized, controlled trial to compare effects of standard versus intensive motor rehabilitation treatment for people with ALS.

Eligible patients are going to be randomly assigned to the Standard or Intensive treatment (controlling for ALSFRSR rates at enrollment, age and site of onset). Randomization ratio is 1:1.

Standard treatment: 2 sessions/week of motor rehabilitation treatment (45 minutes each one) for 10 weeks for a total of 20 sessions. The program consists of exercises for aerobic endurance, reinforcement at low load and stretching. At the end of the 20 sessions patient and caregiver are going to continue activity with supervision through regular follow up.

Intensive treatment is characterized by an increased volume of the above mentioned exercises: 5 sessions/week (45 minutes each one) for 10 weeks for a total of 50 sessions. At the end of the 50 sessions patient and caregiver are going to continue activity with supervision through regular follow up.

Collection and analysis of data

Recruitment: during the first 18 months of the study. Outcome measures: evaluated at T0-T3-T6-T9-T12-T15-T18-T21-T24. Rating scales will be administered by a neurologist in singe blind method with respect to the treatment.

Data collection will be done through an ad hoc Case Report Form and entered into a database on a dedicated website.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of possible, probable or definite ALS according to the Revised El Escorial Criteria
* Time from diagnosis <18 months at screening.
* Forced vital capacity (FVC)> 50% at screening
* Written informed consent

Patients will be required to take the full dose of Riluzole, but not assuming Riluzole do not constitute a criterion for exclusion.

Exclusion Criteria:

* Enrolment in any other clinical trial in the three months prior to screening
* Tracheostomy or NIV for> 23h/day for 14 consecutive days at screening.
* Diagnosis of severe neurodegenerative diseases in addition to the ALS
* Diagnosis of severe heart disease, current neoplasia, any unstable medical condition that contraindicates an intensive rehabilitation treatment
* State of pregnancy or breastfeeding
* Residency outside Emilia-Romagna Region
* Lack of multidisciplinary follow-up

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in ALSFRS R | 12 months

SECONDARY OUTCOMES:
Rate of complications related to the disease: pressure sores, hospitalizations, infections | 12 months
Perceived quality of care | 12 months
Tracheostomy free survival | 12 months
Time to supporting procedures (NIV and PEG) | 12 months
Respiratory function: measured by FVC | 12 months
Quality of Life: measured by McGill and ALSAQ40 scales | 12 months
Disease symptoms (fatigue) measured with FSS | 12 months
Depression measured by Beck Inventory Scale | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marco Vinceti, MD, Study Chair — Public Health Department, University of Modena and Reggio Emilia (IT)
Locations (3):
- Italy (3):
  - Department of Neuroscience, S. Anna Hospital, Ferrara
  - Department of Neuroscience, S.Agostino-Estense Hospital, Modena
  - Department of Neuroscience, IRCCS Arcispedale Santa Maria Nuova, Reggio Emilia